CLINICAL TRIAL: NCT05273385
Title: Efficacy of the Nanodropper Device on Intraocular Pressure in Patients With Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Nanodropper, Inc. (Industry); Icare Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-32530
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma; Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study personnel who will evaluate the IOP and economic endpoints will be blinded to patients' assigned dispenser types for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Nanodropper (Experimental): Participants will receive the Nanodropper with instructions and attend clinic visits at baseline, 1, and 3 months. Participants will administer their eye drops using the Nanodropper.
  Interventions: Device: Nanodropper
- Standard of Care Dropper (No Intervention): Participants will receive standard of care eye dropper with instructions and attend clinic visits at baseline, 1, and 3 months. Participants will administer their eye drops using the standard of care eye dropper.

INTERVENTIONS:
Device: Nanodropper — Device to apply liquid medication to eyes
  Arms: Nanodropper

SUMMARY:
Glaucoma is the leading cause of irreversible blindness worldwide. Previous studies demonstrate that smaller eye drops used in the treatment of glaucoma are just as efficacious as their larger counterparts. The proposed study hopes to demonstrate the non-inferiority of using Nanodropper to lower intraoccular pressure (IOP) in glaucoma patients compared to standard of care eye drops.

DETAILED DESCRIPTION:
The proposed study strives to demonstrate the non-inferiority of using Nanodropper to lower IOP in glaucoma patients compared to standard of care (SOC) eye drops in a randomized trial.

Primary Aim: Demonstrate non-inferiority of using Nanodropper to lower IOP compared to standard of care eye drops in glaucoma patients.

Stable glaucoma participants and ocular hypertension participants of ages 18+ will be randomized to either use Nanodropper for eye drop administration in both eyes OR administer drops regularly (standard of care) in both eyes. Participants will be followed-up at 1 month and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Diagnosis of open-angle glaucoma (OAG) or ocular hypertension (OHT)
3. Use of prostaglandin analogue (PGA) eye drop
4. Stable disease status (no visual field loss progression or increase in IOP-lowering medications in the last 6 months)

Exclusion Criteria:

1. Uncontrolled glaucoma
2. Have had eye surgery (including laser procedures) within the past six months
3. Have a diagnosis of acute angle-closure glaucoma and/or other retinal diseases
4. Use of non-PGA class of IOP-lowering medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) at Baseline | At Baseline
  IOP measurement of the eye will be collected at the baseline visit using routine methods including Goldman applanation tonometry and pneumotonometer.
Intraocular pressure (IOP) at Month 1 | 1 month
  IOP measurement of the eye will be collected at the Month 1 visit using routine methods including Goldman applanation tonometry and pneumotonometer.
Intraocular pressure (IOP) at Month 3 | 3 months
  IOP measurement of the eye will be collected at the month 3 visit using routine methods including Goldman applanation tonometry and pneumotonometer.

SECONDARY OUTCOMES:
Survey | 3 months
  The following open-ended questions will be administered to participants randomized to the Nanodropper group at the end of the 3-month study.
  1. Would you consider using the Nanodropper for your regular eye drop use in the future? (yes/no)
  2. Did you find the Nanodropper easy to use? (yes/no)
  3. Did using the Nanodropper cause more irritation compared to normal eye drop bottles? (yes/no)
Conjunctival Grading at Baseline | At baseline
  Conjunctival grading will be performed by a masked ophthalmologist at the baseline study visit. Grading will be performed with redness graded on a scale of 0-100 using the bulbar redness 5-picture validated scale.
Conjunctival Grading at Month 3 | 3 months
  Conjunctival grading will be performed by a masked ophthalmologist the 3 month study visit. Grading will be performed with redness graded on a scale of 0-100 using the bulbar redness grading 5-picture validated scale.

CONTACTS AND LOCATIONS:
Overall Officials: Julius Oatts, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification(text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. For individual participant data meta-analysis.